CLINICAL TRIAL: NCT01041911
Title: Double-blind, Randomized, Placebo-controlled, Dose Response Study to Evaluate the Safety and Efficacy of Three Doses of Euphorbia Prostrata Dry Extract Tablets in Patients of Hemorrhoids
Brief Title: To Evaluate the Dose Response of 3 Doses of Euphorbia Prostrata in Patients With First and Second Degree Hemorrhoids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Panacea Biotec Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBL/CR/0102008/CT
Record Dates: First submitted 2009-12-31; First posted 2010-01-01 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Euphorbia 50 mg (Active Comparator): This arm subjects will be given 50 mg Euphorbia prostrata
  Interventions: Drug: Euphorbia tablets
- Euphorbia 100 mg (Active Comparator): In this arm subjects will be given 100 mg Euphorbia
  Interventions: Drug: Euphorbia tablets
- Euphorbia 200 mg (Active Comparator): In this arm subject will be given 200 mg Euphorbia tablets
  Interventions: Drug: Euphorbia tablets
- Placebo (Placebo Comparator): In this arm subjects will be given placebo tablets
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: Euphorbia tablets — 50 mg, tablet, once daily, 14 days
  Other Names: To be confirmed later
  Arms: Euphorbia 50 mg
Drug: Euphorbia tablets — 100 mg, tablet, once daily, 14 days
  Other Names: To be confirmed later
  Arms: Euphorbia 100 mg
Drug: Euphorbia tablets — 200 mg, tablet, 2 tablets of 100 mg Euphorbia prostrata, 14 days
  Other Names: To be confirmed later
  Arms: Euphorbia 200 mg
Drug: Placebo tablets — placebo, tablet, once daily, 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safe and efficacious dose of Euphorbia prostrata for control of per rectal bleeding in patients with first and second degree hemorrhoids.

DETAILED DESCRIPTION:
Hemorrhoidal disease is a common entity in the general population and in clinical practice. The basic pathological factor in hemorrhoids is the dilation of the anorectal venous plexuses. In the acute bleeding of internal hemorrhoids, one of the pathogenic processes implicated is the stagnation and stasis of blood in the vascular plexuses of the prolapsed anal cushions. Euphorbia prostrata extract is found to have antihemorrhoidal activity and is useful in ameliorating signs and symptoms associated with hemorrhoids.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects who are able to understand nature, significance and scope of the clinical trial and express their will accordingly and agreeing to participate in the study by giving written informed consent.
* Male or female subjects, at least 18 years of age with a diagnosis of internal hemorrhoids (first and second degree) confirmed by proctoscopic examination and suffering from an uncomplicated and untreated acute attack (defined as acute onset of per rectal bleeding within 3 days of inclusion into the study, with at least one of the symptoms viz. pain, tenesmus, pruritus and anal discharge).
* Except internal hemorrhoids (first and second degree), the subjects are judged to be in good general health, based on medical history, physical examination, and laboratory screening tests.

Exclusion Criteria:

* Pregnant and lactating women and women in post-partum period of up to 6 weeks.
* Women of child bearing potential who do not agree to remain abstinent or use medically acceptable methods of contraception during the study therapy and for 4 weeks after the end of study therapy.
* Subjects who have been previously enrolled in a study involving E. prostrata Dry Extract
* Subjects with a history of permanent anal prolapse and/or anal fistula
* Subjects with associated anal fissures and/or infective anal pathology.
* Subjects with previous history of surgery for anorectal disease (within 5 years) or any other procedures (including but not limited to injection sclerotherapy, rubber band ligation, photocoagulation, cryotherapy etc) within 2 year of enrolment into the trial.
* Subjects who, in the opinion of the investigator, are mentally incapacitated such that informed consent cannot be obtained.
* Subjects with clinically significant co-morbid condition that in the opinion of the investigator could affect the efficacy and safety outcome of the study.
* Subjects with clinically significant laboratory values for hemoglobin, total leukocyte count, differential count, bleeding time, clotting time, PT/INR, aPTT/control, platelet count, SGOT, SGPT, alkaline phosphatase, total bilirubin, random blood sugar, serum cholesterol, blood urea, serum creatinine and urine routine and microscopic examination.
* Treatment with any of the following at inclusion or in the previous one month venotropic, anticoagulant, and anti platelet agent. Subjects on aspirin up to 160 mg for cardiovascular indication will not be excluded from the trial.
* Treatment with any of the following at inclusion or in the previous one week anti-inflammatory and analgesic agent.
* Other chronic medications not being used at a stable dosage for at least 2 weeks.
* Subjects who are current users of illicit drugs including "recreational use" or with a history of drug abuse within the past 5 years.
* Subjects who have donated a unit of blood or plasma or participated in another clinical study with an investigational agent within the last 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in each treatment group achieving cessation of per rectal bleeding as assessed by the subject | 14 day of treatment

SECONDARY OUTCOMES:
Proportion of subjects in each treatment group without recurrence of bleeding | 14 days post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dr P N Agarwal, Principal Investigator — Maulana Azad Medical College, New Delhi; Dr Girish Bakshi, Principal Investigator — Grant Medical College, Mumbai; Dr T Durganna, Principal Investigator — Bangalore Medical College, Bangalore; Dr Saiprasad Donga, Principal Investigator — Sahil Hospital, Tawdw Niwas, 1st Floor Khopat, Thane; Dr Vaibhav Lokhande, Principal Investigator — Nath Hospital, Golden Heaven Society, Opp Janta Sahakari Bank, Khopat, Thane; Dr P S Sarangi, Principal Investigator — Deen Dayal Upadhyay Hospital, Hari Nagar, New Delhi
Locations (6):
- India (6):
  - Bangalore Medical College, Bangalore, Karnakata
  - Grant Medical College, Mumbai, Maharashtra
  - Nath Hospital, Golden Heaven Society, Opp Janta Sahakari Bank,, Thane, Maharashtra
  - Sahil Hospital, Tawdw Niwas, 1st Floor Khopat, Thane (W), Thane, Maharashtra
  - Maulana Azad Medical College, New Delhi, National Capital Territory of Delhi
  - Deen Dayal Upadhyay Hospital, Hari Nagar, New Delhi, New Delhi, National Capital Territory of Delhi